CLINICAL TRIAL: NCT00062101
Title: A Phase II Study of OSI 774 (IND Number 63383) in Combination With Celecoxib (Celebrex, Pharmacia) as Second-Line Therapy in Advanced Non-Small Cell Lung Cancer
Brief Title: Erlotinib and Celecoxib in Treating Patients With Stage IIIB or Stage IV Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02720; LUNG 2002-01; NCI-5416; CDR0000304495
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Celecoxib

ARMS (2):
- Group I (erlotinib hydrochloride, celecoxib) (Experimental): Patients receive oral erlotinib once daily and oral celecoxib twice daily.
  Interventions: Drug: erlotinib hydrochloride; Drug: celecoxib; Other: laboratory biomarker analysis
- Group II (erlotinib hydrochloride) (Experimental): Patients receive erlotinib as in group 1.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally (PO)
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: celecoxib — Given PO
  Other Names: Celebrex; SC-58635
  Arms: Group I (erlotinib hydrochloride, celecoxib)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving erlotinib together with celecoxib works in treating patients with recurrent stage IIIB or stage IV non-small cell lung cancer. Erlotinib and celecoxib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Celecoxib may slow the growth of a tumor by stopping blood flow to the tumor. Combining erlotinib with celecoxib may kill more tumor cells.

.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate of patients with stage IIIB or IV recurrent non-small cell lung cancer treated with erlotinib and celecoxib as second-line therapy.

SECONDARY OBJECTIVES:

I. Determine the time to progression in patients treated with this regimen. II. Determine the survival duration of patients treated with this regimen. III. Determine the toxicity of this regimen in these patients. IV. Correlate the expression of epidermal growth factor receptor and cyclooxygenase-2 in tumor specimens with response, time to progression, and survival in patients treated with this regimen.

OUTLINE: Patients are assigned to 1 of 2 treatment groups.

Group 1: Patients receive oral erlotinib once daily and oral celecoxib twice daily.

Group 2: Patients receive erlotinib as in group 1.

Treatment in both groups continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 40-80 patients will be accrued for this study within 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage IIIB (malignant pleural effusion only) or IV
* Recurrent disease that has progressed after 1 or 2 prior chemotherapy regimens (platinum- or nonplatinum-based)
* At least 1 unidimensionally measurable lesion*

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* Must have tissue specimen available for assays
* No brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST/ALT no greater than 2.5 times upper normal limit (ULN)
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No prior abnormalities of the cornea (e.g., dry eye syndrome or Sjögren's syndrome)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
* No abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)
* Able to ingest oral medication
* No requirement for IV alimentation
* No history of peptic ulcer disease
* No active gastrointestinal ulcers
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No significant traumatic injury within the past 21 days
* No psychiatric illness or social situation that would preclude study compliance
* No prior allergic reactions to sulfonamides, aspirin, and other nonsteroidal anti-inflammatory drugs
* No prior monoclonal antibodies to epidermal growth factor receptor (EGFR)
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No concurrent chemotherapy
* No concurrent glucocorticoids
* More than 4 weeks since prior radiotherapy and recovered
* More than 21 days since prior major surgery
* No prior surgery affecting absorption
* No prior EGFR-specific tyrosine kinases
* No concurrent anticonvulsants
* No other concurrent investigational agents
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent antacids
* No concurrent administration of any of the following drugs:

  * Amiodarone
  * Chloramphenicol
  * Cimetidine
  * Fluvoxamine
  * Omeprazole
  * Zafirlukast
  * Clopidogrel
  * Cotrimoxazole
  * Disulfiram
  * Fluconazole
  * Fluoxetine
  * Fluvastatin
  * Fluvoxamine
  * Isoniazid
  * Itraconazole
  * Ketoconazole
  * Leflunomide
  * Metronidazole
  * Modafinil
  * Paroxetine
  * Phenylbutazone
  * Sertraline
  * Ticlopidine
  * Valproic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-01; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Response rate according to the Response Evaluation Criteria in Solid Tumors (RECIST) | From the start of treatment until disease progression/recurrence, assessed up to 5 years

SECONDARY OUTCOMES:
Time to progression | Interval between start of treatment with erlotinib hydrochloride and celecoxib and the date on which progressive disease, assessed up to 5 years
  Will be analyzed by calculating Kaplan Meier curves and estimating medians and 95% confidence intervals using the method of Brookmeyer and Crowley.
Overall survival | Up to 5 years
  Will be analyzed by calculating Kaplan Meier curves and estimating medians and 95% confidence intervals using the method of Brookmeyer and Crowley.
Relationship between measures of treatment efficacy and EGFR and COX-2 levels | Up to 5 years
Toxicity as assessed by NCI Common Toxicity Criteria (CTC) version 2.0 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bonomi, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States